CLINICAL TRIAL: NCT01971034
Title: A Prospective Study to Evaluate the Combination of Metformin With Paclitaxel in the Treatment of Patients With Advanced Pancreatic Cancer After Gemcitabine Failure.
Brief Title: Treatment of Patients With Advanced Pancreatic Cancer After Gemcitabine Failure.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 96/2010
Record Dates: First submitted 2013-09-06; First posted 2013-10-28 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Adenocarcinoma Advanced or Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Paclitaxel; Metformin

ARMS (1):
- Paclitaxel and Metformin (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Metformin

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m2, IV, Day 1, Day 8 and Day 15.
Drug: Metformin — 850mg, PO, every 8 hours, daily.

SUMMARY:
In Brazil pancreatic adenocarcinoma represents 2% of tumors, and 4% mortality being an uncommon disease, however very aggressive.Only 20% of cases are indicated for curative surgery, of which only 20% are alive within 5 years. For locally, advanced or metastatic disease, since 1997, single chemotherapy with gemcitabine is the standard treatment for first line, with survival around 6 months approximately.There is no standard treatment regimen for second-line, however Paclitaxel demonstrated effect on second-line phase II study. Metformin is an oral hypoglycemic drug used for treatment of diabetes mellitus. There is a growing number of preclinical studies which show antitumor effect against pancreatic adenocarcinoma, probably due to the effect of anti-insulin growth factor (IGF-1). This study will add metformin to standard treatment for second line of locally advanced or metastatic pancreatic adenocarcinoma in ICESP previously treated with gemcitabine. The objective is to evaluate whether metformin improves the efficacy of the standard treatment with paclitaxel by clinical and radiological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic advanced or metastatic adenocarcinoma histologically confirmed.
* Previously treatment with gemcitabine as adjuvant or metastatic disease.
* Clinical or radiological evidence of disease progression, determined by physician. Is not mandatory RECIST (Response Evaluation Criteria in Solid Tumors) evaluation to determine the progression of disease before the study inclusion.
* Patient with intolerance to gemcitabine, even without disease progression, are also eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* At least 10 weeks of life expectation.
* Adequate organ function defined as:

  * Serum AST (aspartate aminotransferase) and ALT (alanine aminotransferase)≤ 2.5 × ULN (upper normal limit)
  * Total Bilirubin ≤ 2,0 x ULN
  * Absolute neutrophil count ≥ 1,500/ mm3
  * Platelets ≥100.000/ mm3
  * Hemoglobin ≥ 8,0 g/dl
  * Serum Creatinine ≤ 1,5 ULN and clearance of creatinine estimated (Cockcroft- Gault) ≥ 50 ml/min
* Signed written informed consent.

Exclusion Criteria:

* Major surgical procedure within 4 weeks of the beginning of the treatment.
* History of serious clinical or psychiatric disease.
* Symptomatic hypoglycemia at the screening visit.
* Target lesion radiotherapy within 4 weeks of the beginning of the treatment.
* Treatment with any anti-cancer investigational drug.
* Treatment with any IGF-I or IGFR-I
* Treatment with metformin within 12 months prior to commencing study treatment
* For female patients, current pregnancy and/or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Radiologic control of disease | Every 8 weeks from the date of first dose of treatment until disease progression.
  The radiologic image will be analyzed by RECIST 1.0 criteria.

SECONDARY OUTCOMES:
Time to progression. | Every 8 weeks from the date of first dose of treatment until disease progression.
  Thorax and abdominal computerized tomography and Ca 19.9 tumor marker dosage every 8 weeks until disease progression.
To estimate the biochemical response through the measurement of serum CA19.9 levels. | From the date of first dose of treatment until disease progression.
To evaluate the clinical benefits | Every 4 weeks during the treatment period until disease progression.
  Will be evaluate:
  * ECOG
  * Treatment with opioids
  * Pain
  * Weight

CONTACTS AND LOCATIONS:
Overall Officials: Rachel SP Riechelmann, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.icesp.org.br